CLINICAL TRIAL: NCT05546021
Title: Influence of Nociception Level Monitor (NOL) During Guided Analgesic Delivery in Breast Surgeries on the Perioperative Course, Quality of Recovery and Hospital Stay
Brief Title: Nociception Level Monitor (NOL) During Guided Analgesic Delivery in Breast Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SHS-An-1-2022
Record Dates: First submitted 2022-08-30; First posted 2022-09-19 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Anesthesia; Adverse Effect; Breast Cancer
Keywords: nociception level monitor
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOL monitor (Active Comparator): Patients will receive opioids as per the guidance of a nociception level monitor (NOL)
  Interventions: Procedure: NOL monitor
- Standard care (No Intervention): Patients will be treated as per the department´s standard protocol.

INTERVENTIONS:
Procedure: NOL monitor — NOL technology uses a multiparameter-based sensor platform, and advanced algorithm, to continuous monitor Autonomic Nervous System (ANS) functions. NOL reflects a patient's nociceptive state and analgesic effect, helping to optimize the administration of systemic and/or regional analgesics and avoiding overdose or underuse of these drugs.
  The nociception level is a multiparameter monitor that combines information from the finger photoplethysmogram amplitude, skin conductance, skin conductance fluctuation, heart rate, heart rate variability, and their time derivatives into one index ranging from 0 (absence of noxious stimulation) to 100 (severe noxious stimulation). The nociception level is a composite score derived from a set of physiologic variables (i.e., peripheral effectors of the autonomous nervous system): heart rate, heart rate variability, the amplitude of the photoplethysmogram, skin conductance, skin conductance variability, and the time derivatives of these variables.
  Arms: NOL monitor

SUMMARY:
To assess if perioperative consumption of opioids can be optimized with the assistance of a Nociception Level (NOL) monitor in breast surgery patients receiving pectoral and parasternal nerve blocks as supplementation to general anaesthesia.

Hypothesis:

1. NOL monitor guidance optimizes perioperative analgesic consumption and postoperative length of stay and offers a better quality of recovery in breast surgery.
2. Intraoperative NOL monitoring can detect the efficacy of pectoralis and parasternal nerve blocks.
3. Incidence of persistent neuropathic pain after breast cancer surgery is lower in patients receiving lower doses of perioperative opioids.

DETAILED DESCRIPTION:
Optimal perioperative pain management is important not only for patient satisfaction but also for hemodynamic stability and effective restitution. Despite being the principal element of anaesthesia, analgesia delivery has long been based on non-objective surrogate parameters such as blood pressure and heart rate. This may lead to hemodynamic inconsistency, poor restitution and patient dissatisfaction, which are some of the observed challenges. In that context, there has long been a search for a monitor which can guide the meticulous administration of analgesics. Recently, a nociception level monitor (NOL) based on an advanced software algorithm was developed using multiple physiological parameters. It offers an objective number (NOL Index) which relates to the level of intra-operative pain. NOL technology has been validated and found superior to existing pain indicators in peer-reviewed publications. With the availability of NOL monitors, a meticulous adjustment in the administration of opioids became a possibility. Therefore, the investigators are planning a randomised study to investigate if opioid consumption can be reduced and if immediate and long-term postoperative complications can be minimised.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists (ASA) class I-IV patients scheduled for an elective mastectomy with or without axillary resection

Exclusion Criteria:

* Inability to give consent,
* atrial fibrillation,
* local anesthetic allergy,
* lumpectomy converted to Mastectomy.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Peroperative Remifentanil consumption | during the surgery
  ( peroperative, mg)
Peroperative Morphine consumption | during the surgery
  (peroperative, mg)

SECONDARY OUTCOMES:
Postoperative Maximum pain score | immediately after the surgery
  measured using numerical rating scale (NRS) (0-10). The score can vary between 0 and 10 by which 0 means no pain and 10 equals the worst possible pain.
Post-operative opioid consumption | immediately after the surgery
  Morphine, mg
Eligible time to discharge | immediately after the surgery
  Time in the post anaesthesia care unit based on a post anaesthesia care score scheme derived from objective vital parameters (Minutes)
Length of hospital stay | From admission to discharge, up to 72 hours
  Hours
Incidence of post-operative nausea and vomiting | immediately after the surgery
  Number of patients with post-operative nausea and vomiting
Requirement for additional antiemetic drugs | immediately after the surgery
  Number 1-3
Persistent neuropathic pain after breast cancer surgery | up to 3 months after surgery
  Number of patients experiencing pain due to breast cancer surgery measured using numerical rating scale (NRS) (0-10). The score can vary between 0 and 10 by which 0 means no pain and 10 equals the worst possible pain.
Length of time in recovery room | immediately after surgery
  minutes

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Prabhakar Bhavsar, Principal Investigator — University of Hospital of Southern Denmark - Aabenraa
Locations (1):
- Sygehus Soenderjylland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edry R, Recea V, Dikust Y, Sessler DI. Preliminary Intraoperative Validation of the Nociception Level Index: A Noninvasive Nociception Monitor. Anesthesiology. 2016 Jul;125(1):193-203. doi: 10.1097/ALN.0000000000001130. PMID 27171828
- [Background] Martini CH, Boon M, Broens SJ, Hekkelman EF, Oudhoff LA, Buddeke AW, Dahan A. Ability of the nociception level, a multiparameter composite of autonomic signals, to detect noxious stimuli during propofol-remifentanil anesthesia. Anesthesiology. 2015 Sep;123(3):524-34. doi: 10.1097/ALN.0000000000000757. PMID 26154185
- [Background] Stockle PA, Julien M, Issa R, Decary E, Brulotte V, Drolet P, Henri M, Poirier M, Latulippe JF, Dorais M, Verdonck O, Fortier LP, Richebe P. Validation of the PMD100 and its NOL Index to detect nociception at different infusion regimen of remifentanil in patients under general anesthesia. Minerva Anestesiol. 2018 Oct;84(10):1160-1168. doi: 10.23736/S0375-9393.18.12720-9. Epub 2018 May 14. PMID 29756750
- [Background] Malachauskiene L, Bhavsar R, Bakke S, Keller J, Bhavsar S, Luy AM, Strom T. Influence of Nociception Level Monitor (NOL)-Guided Analgesic Delivery on Perioperative Course in Breast Surgeries: A Randomized Controlled Trial. Medicina (Kaunas). 2024 Nov 22;60(12):1921. doi: 10.3390/medicina60121921. PMID 39768803